CLINICAL TRIAL: NCT06149364
Title: Cost-effectiveness and Impact of a Workplace-based Intervention to Reduce Occupational Sitting Time Among Office-based Workers: a Randomized Controlled Trial
Brief Title: Cost-effectiveness, Impact of a Workplace-based Intervention to Reduce Occupational Sitting Time in Office-based Workers
Acronym: ISKE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Principal Investigator, Sanaz Akhavan Rad, Doctoral Researcher, University of Helsinki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S1371
Record Dates: First submitted 2023-11-15; First posted 2023-11-29 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity; Sedentary Behavior; Occupational Diseases; Physical Activity
Keywords: Cost-effectiveness; Economic evaluation; Randomized control trial; Sitting time; Workplace; Office workers; Productivity; Absenteeism; RCT
MeSH Terms: conditions — Sedentary Behavior; Occupational Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Experimental): Control - usual practice; participants in this arm will be informed that the project is aimed at an economic evaluation of costs associated with usual patterns of office-based routines among desk-based workers. The measurements for both CG and IG will be taken at four times (baseline, 3 months, 6 months, and 12 months).
  Interventions: Behavioral: ISKE

INTERVENTIONS:
Behavioral: ISKE — The intervention will consist of an e-health software Programme that we have named "Istumisen Keskeyttäminen (ISKE)" will be installed on the desktop of participants.
  Functionality of the software: the primary purpose of the software is to remind users (basically office-based workers) to take a break on a regular basis (recommended time 30 minutes).
  At the end of the workday, the software provides information on the number of breaks taken and how long each lasted. The user will also have access to such information.
  What happens during the prompted break: once the software prompts the user to take a break, she/he can click the Continue button to proceed with the break. The software will include activities that are suggested for the user to do during break. After the break, the record of the time (duration of the break, and when the break was taken) can be taken.

SUMMARY:
The purpose of this study is to examine the impact and cost effectiveness of a workplace-based intervention aimed at reducing prolonged occupational sitting among office-based workers. The study will be conducted in three phases. Phase I: is an Integrative review on economic evaluations of workplace-based interventions for reducing occupational sitting time. Phase II: is a secondary analysis of register data within the Northern Finland Birth Cohort 1966 (NFBC-1966). This is aimed at evaluating the association between prolonged sitting time with societal and/or organization economic perspective across different occupational categories at midlife. Phase III will be a Randomized Control Trial (RCT) of an office-based intervention designed to reduce prolonged occupational sitting time. The sample for the RCT will be 140 office-based workers - 70 participants will be enrolled in the control group whilst 70 participants will be enrolled within the intervention group. The study will be conducted from 2021 to 2025. An article-based dissertation will be completed at the end of the study, this will be mainly based on four articles that will be published in international peer reviewed journals.

DETAILED DESCRIPTION:
In office-based work environments, prolonged durations of sitting are the commonest form of daily sedentary behavior within which the most sitting time (47.2% of total daily sitting time). Sedentary behavior has been associated with up to 1.5 ¬3% of the total direct health, about US$ 13.7 billion incurred in production loss costs, and 13.4 million due to disability-adjusted life years globally. In Finland, physical inactivity and sedentary behavior resulted in a total healthcare cost of €3.2 billion due to low physical activity and €1.5 billion due to high sedentary behavior. Sustaining healthy and productive workers is a substantial goal of the European labor policy thus, there is need for workplace-based interventions to promote healthy sitting at workplaces.

Objectives of the Study

General objective:

The purpose of this study is to examine the impact and cost-effectiveness of a workplace intervention for reducing prolonged occupational sitting among office-based workers.

Specific objectives:

(i) To assess the existing evidence on economic evaluation of workplace interventions aimed at reducing prolonged occupational sitting among office-based workers (Phase I).

(ii) To determine the societal and/or organizational cost-perspective association with sitting time within various occupational categories (Phase II) (iii) To examine the impact and cost-effectiveness of a workplace physical activity intervention aimed at reducing prolonged occupational sitting using a randomized controlled design (Phase III) Methods

Study design and study population:

The study will be conducted in three phases corresponding to distinct objectives, designs, data collection and analysis approaches.

Phase I The search was conducted in 11 databases, including PubMed, Scopus, PsychINFO, NHS-EED, Cumulative Index to Nursing and Allied Health Literature (CINAHL), ProQuest, Cochrane library, Sportdiscus, Research Paper in Economics (RePeC), the International Health Economic Association (IHEA) and EconLit. Phase II: Data will be obtained from the Northern Finland Birth Cohort 1966 (NFBC-1966) and data collected from the Finland´s national registers on direct and indirect costs related to the use of health care services and absence from work. Data will be extracted on: health care utilization, informal care, productivity losses (sickness absenteeism: paid and unpaid work, presenteeism) and lost productivity cost.

Phase III The study design: The sub-study is designed as a non-blinded randomized control trial (RCT) among office workers. The sub-study is planned to be executed within 12-months. The data points will be at baseline, 3 months, 6 months and at 12 months. The CONSORT guidelines (Moher et al., 2010) will be adopted for this study.

Sample size estimation based on power: The sample size was computed based on power analysis. Considering that our primary outcome is a continuous variable, and we wish to have a 0.90 power of our intervention - a similar RCT had a relatively higher power (0.91) among office workers; mean reduction in sitting time for group 1 (266.01 minutes/workday) and mean group 2 (78.26 minutes/workday), an estimated sample of 70 participants per group will be required with an enrollment ratio of 1:1 and Beta of 0.1 at 0.05. An RCT provides the strongest evidence of any design that a given intervention has a postulated effectiveness.

Participants recruitment: The accessible population of office-based workers from the University of Oulu will be approached through that occupational care provider on a rolling basis. Further information will be provided to them through their occupational health organization (Mehiläinen) at Oulu University. Information about the invitation and participation in the study is known to the researchers and the person in charge of the occupational health care study, but not to the employer.

At the time of recruitment, potential participants will be provided information via meetings (physical or online), phone calls, short messaging service or emails. The target is to recruit 140 participants (e.g., 70 participants in the control group and 70 participants in the experimental group).

Initially, through the designated contact person within Mehiläinen, the researcher will provide information about the study using an information leaflet via email to eligible participants The process of providing information will be supplemented by clarifications from the researcher on issues that may require further explanation. After having time enough to read the information on the study, those that accept to participate in the study will be randomized into the control group or the experimental group. Randomization will be conducted by generating random numbers (www.randomization.com). Before the intervention, participants recruited in the experimental group will undergo an orientation session (physical or online). This will be a 15- minute educational session on prolonged sitting, general instructions on performing appropriate workplace physical activity, and how to use the software and accelerometer and illustrations about how the passive prompting e-health software works will be conducted. The prompting software, accelerometer and tools will be distributed to participants at the same time.

The intervention:

Control - usual practice; participants in this arm will be informed that the project is aimed at an economic evaluation of costs associated with usual patterns of office-based routines among desk-based workers. The measurements for both CG and IG will be taken at four times (baseline, 3 months, 6 months, and 12 months).

The experimental group will receive a multicomponent intervention. The intervention will consist of an e-health software Programme that we have named "Istumisen Keskeyttäminen (ISKE)" will be installed on the desktop of participants.

Functionality of the software: the primary purpose of the software is to remind users (basically office-based workers) to take a break on a regular basis (recommended time 30 minutes).

The initial features of the software have been specifically designed for this study. When the participant opens the software, a Setup Assistant window will appear allowing the user to register and customize the nature of the alerts/breaks. The setup window also has a suggested mode - "Standard" break will default to every 30 minutes from the time when the user starts the day.

At the end of the workday, the software provides information on the number of breaks taken and how long each lasted. The user will also have access to such information.

What happens during the prompted break: once the software prompts the user to take a break, she/he can click the Continue button to proceed with the break. The software will include activities that are suggested for the user to do during break. It is possible to include a list of examples of exercises that can be done within the office based.

After the break, the record of the time (duration of the break, and when the break was taken) can be taken.

Progress of the break bar:

While in a break, a progress bar shows how long till the break is over.

Postpone option:

The break can also be postponed via the Postpone Button. It allows the user to skip taking the break with options to remind the user to take the break in for example: 5 minutes later or 10 minutes. The software also provides information on the total number of times you have postponed.

Rewarding the users:

virtual badges are also included in the software - they are aimed to reward and sustain motivation to use the software. These will be based on their extent of use of the software and in turn their activity time/ sitting time. For example, frequent break followers are rewarded a badge more frequently. These virtual badges are based on activity level of users anonymously. virtual reward-related information is not collected in the research material but is intended to motivate the participants.

The software does not collect any data from the users´ computer. The software has been designed to generate user tokens (App identification). The Administrator (researcher) will input basic user information, generates tokens and send it to the user. This way, we simplify the user management process, because we don't need user info username (for purpose of privacy, this doesn't require the person to use their real names), password handling and resetting functions at all in the app.designed by Finnish company developer based on suggested features of researchers in a simple way aimed to easily use and reduce distraction of users.

Before the intervention, participants recruited in the experimental group will undergo an orientation session. The session will be physical or online. During the orientation session, participants will be given a 15- minute educational session on the negative health effects associated with prolonged sitting, general instructions on performing appropriate workplace physical activity, during this session, illustrations about how the passive prompting e-health software works and how to use an accelerometer will be conducted. Participants will be asked to wear the accelerometer (ActivePal) for 14 days during workdays hours in the thigh.

How the data is collected:

The hypothesis of the third sub-study is that the intervention will reduce sitting time. Consequently, over the long term, it will lead to reduction in absenteeism, presenteeism, enhance Quality adjusted life year (QALY) and reduce exhaustion at work.

Assessments will be done at baseline, 3 months, 6 months, and 12 months. Data from activity monitoring, and a self-administered questionnaires will be used.

The research materials and instruments will be distributed online via email to eligible participants during phase III. These will include the information leaflet, data protection statement, consent form and tools.

Measuring sitting time and physical activity: Physical activity will be objectively measured with the ActivePal accelerometer (PAL technologies LTD, Glasgow, UK). This is a thigh-worn, tri-axial accelerometer. The accelerometer was chosen because it is easy to use, discrete and can differentiate between sitting, standing, and stepping in varying postural transitions (Boudet et al., 2019). Participants will be asked to wear the monitors for at least 14 days during workdays hours. The participants will then give the accelerometer to the researcher, data recorded on them will be downloaded and analyses.

Data protection: Handling of personal data will be done according to the principles of the EU General Data Protection Regulation (EU 679/2016) and Data Protection Act. Strategies will be implemented to ensure that research is not harmful to the employment relationship of the participants. Ideally, the employee's supervisor will have no contact with the employee during recruitment, enrollment, assessment of outcomes, nor will the supervisor have access to the employee's identified data and sample.

Analysis approaches: Differences in sitting time per 8 working hours based on the accelerometer within the control group and the experimental group will be examined. The association of sitting rate and other variables (absenteeism, presenteeism, QALY, job satisfaction and exhaustion) will be analyzed. Individual level differences within the experimental group will be analyzed with respect to variations in number of breaks taken during the working hours.

Ethical consideration: The current study protocol will be reviewed and approved by the Research Ethics committee of the Faculty of Medicine of the University of Helsinki. Participation in the study will be entirely voluntary and participants will be allowed to exit from the study at any time when they wish to do so. Personal data of the participants will be protected un the European regulation for personal data protection. The Helsinki Declaration on conduct of research involving human subjects will also be followed in this study.

ELIGIBILITY:
Inclusion Criteria:

* working at least six full time hours
* Age of 18-65 years
* Speaking Finnish language
* Having designated access to internet
* Telephone, and a desk within their workplace (home and away from home workplaces will be considered).

Exclusion Criteria:

* Non-ambulatory
* Pregnant
* Those participating in other RCTs
* Those planning relocation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Assessments will be done at baseline, 3 months, 6 months, and 12 months. Data from activity monitoring, and a self-administered questionnaires will be used.
  Physical activity will be objectively measured with the ActivePal accelerometer (PAL technologies LTD, Glasgow, UK). This is a thigh-worn, tri-axial accelerometer. The accelerometer was chosen because it is easy to use, discrete and can differentiate between sitting, standing, and stepping in varying postural transitions. Participants will be asked to wear the monitors for at least 14 days during workdays hours. The participants will then give the accelerometer to the researcher, data recorded on them will be downloaded and analyses.

SECONDARY OUTCOMES:
Cost | Assessments will be done at baseline, 3 months, 6 months, and 12 months
  Costs will be measured using the full cohort data for the control and intervention group including intervention costs, visits to the occupational health care, participant time spent on intervention and estimated work loss costs due to absenteeism/ sickness absence.
Absenteeism | Assessments will be done at baseline, 3 months, 6 months, and 12 months
  Work time missed,will be objectively measured through employer-recorded absence data for the intervention and control participants. Costs according to the reason of absence e.g., sickness leave will be obtained from the occupational health records and the employer.
Presenteeism | Assessments will be done at baseline, 3 months, 6 months, and 12 months
  Impairment at work/ reduced on-the-job effectiveness will be measured with Presenteeism Scale.
Health related quality of life | Assessments will be done at baseline, 3 months, 6 months, and 12 months
  will be measure with the Finnish version of the European Quality of Life with Five Domains (EQ-5D-5L), this questioner has three levels of quality in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Raija Korpelainen, Phd, Study Director — Oulu Deaconess Institute Foundation sr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolu P, Kari JT, Raitanen J, Sievanen H, Tokola K, Havas E, Pehkonen J, Tammelin TH, Pahkala K, Hutri-Kahonen N, Raitakari OT, Vasankari T. Economic burden of low physical activity and high sedentary behaviour in Finland. J Epidemiol Community Health. 2022 Jul;76(7):677-684. doi: 10.1136/jech-2021-217998. Epub 2022 Apr 26. PMID 35473717
- [Background] Akhavan Rad S, Kiwanuka F, Korpelainen R, Torkki P. Evidence base of economic evaluations of workplace-based interventions reducing occupational sitting time: an integrative review. BMJ Open. 2022 Jun 30;12(6):e060139. doi: 10.1136/bmjopen-2021-060139. PMID 35772822
- [Background] Tcymbal A, Andreasyan D, Whiting S, Mikkelsen B, Rakovac I, Breda J. Prevalence of Physical Inactivity and Sedentary Behavior Among Adults in Armenia. Front Public Health. 2020 May 5;8:157. doi: 10.3389/fpubh.2020.00157. eCollection 2020. PMID 32432072
- [Background] Deaton A, Cartwright N. Reflections on Randomized Control Trials. Soc Sci Med. 2018 Aug;210:86-90. doi: 10.1016/j.socscimed.2018.04.046. Epub 2018 Apr 28. No abstract available. PMID 29731150
- [Background] Rollo S, Prapavessis H. A Combined Health Action Process Approach and mHealth Intervention to Increase Non-Sedentary Behaviours in Office-Working Adults-A Randomised Controlled Trial. Appl Psychol Health Well Being. 2020 Nov;12(3):660-686. doi: 10.1111/aphw.12201. Epub 2020 Apr 28. PMID 32342662
- [Background] Styles, B., & Torgerson, C. (2018). Randomised controlled trials (RCTs) in education research-methodological debates, questions, challenges. Educational Research, 60(3), 255-264
- [Background] Vanni KJ, Neupane S, Siukola AE, Karinen HM, Pursio HK, Uitti J, Nygard CH. The Presenteeism Scale as a measure of productivity loss. Occup Med (Lond). 2018 Nov 16;68(8):512-518. doi: 10.1093/occmed/kqy124. PMID 30219891
- See also: ISKE study website — http://www.iskestudy.com/